CLINICAL TRIAL: NCT04013087
Title: Randomized, Double-blind, Parallel, Controlled Study to Evaluate the Safety and Nutritional Adequacy of a New Infant Formula in Healthy Term Infants
Brief Title: Safety and Nutritional Adequacy of a New Infant Formula in Healthy Term Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heilongjiang Feihe Dairy Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18-SM-12-FEIHE-001
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Child Development
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Formula (Experimental): Feihe Stage 1 infant formula
  Interventions: Dietary Supplement: Oral feeding of Feihe Stage 1 infant formula
- Control formula (Active Comparator): A commercially available product with comparable composition but does not contain sn-2 palmitate enriched vegetable oil as an ingredient (regular vegetable oil is used)
  Interventions: Dietary Supplement: Oral feeding of control Stage 1 formula
- Breast feeding (Other): Breast fed of human milk
  Interventions: Dietary Supplement: Breast feeding

INTERVENTIONS:
Dietary Supplement: Oral feeding of Feihe Stage 1 infant formula — Oral feeding of Feihe Stage 1 infant formula for 16 weeks
  Arms: Test Formula
Dietary Supplement: Oral feeding of control Stage 1 formula — Oral feeding of control Stage 1 formula for 16 weeks (A commercially available product with comparable composition but does not contain sn-2 palmitate enriched vegetable oil as an ingredient (regular vegetable oil is used))
  Arms: Control formula
Dietary Supplement: Breast feeding — Breast feeding of human milk for 16 weeks
  Arms: Breast feeding

SUMMARY:
This study is a multicenter, double-blind, randomized, controlled, parallel-designed, prospective study and is intended to evaluate the nutritional adequacy and tolerance of a new study formula compared with a concurrent control formula. Approximately 450 infants will be enrolled from approximately 3 China sites. Of these infants, approximately 300 will be randomized 1:1 to receive an investigational formula or a control formula for 16weeks of feeding. The remaining approximately 150 infants will be enrolled as a breastfeeding reference group. The primary outcome measure is the rate of weight gain in g/day between baseline and 16 weeks in the test group compared to control formula group. Participants will have the option of providing stool samples at 8 weeks and 16 weeks for analysis of microbiota and metabolomics. The study period will be 16 weeks, and all infants in the 2 formula groups will receive formula free of charge for 6 months.

DETAILED DESCRIPTION:
Primary Objective

1) Compare the rate of weight gain (in g/day) between infants receiving an investigational formula and infants receiving a control formula between at baseline (B), B+2 weeks, B+4 weeks, B+8 weeks, B+12 weeks, and B+16 weeks.

Secondary Objectives

1. Compare rate of change in length (mm/day) among infants receiving an investigational formula, infants receiving a control formula, and breastfeeding infants at baseline (B), B+2 weeks, B+4 weeks, B+8 weeks, B+12 weeks, and B+16 weeks.
2. Compare rate of change in head circumference (mm/day) among infants receiving an investigational formula, infants receiving a control formula and breastfeeding infants at baseline (B), B+2 weeks, B+4 weeks, B+8 weeks, B+12 weeks, and B+16 weeks.
3. Evaluate and compare achieved body weight, length, and head circumference at each visit and after 16 weeks.
4. Evaluate plotted raw growth data on World Health Organization standard growth charts.1
5. Compare the types and incidence of adverse events among infants receiving an investigational formula, infants receiving a control formula, and breastfeeding infants.
6. Compare average daily intake of formula between infants receiving an investigational formula and infants receiving a control formula.
7. Compare parents' and physician's assessment of formula tolerance among infants receiving an investigational formula, infants receiving a control formula, and breastfeeding infants.
8. Compare counts of Bifidobacteria and Lactobacillus species in stools of infants receiving an investigational formula, infants receiving a control formula, and breastfeeding infants.
9. Compare stool short-chain fatty acid metabolites (including total SCFAs, acetic, propionic, n-butyric, iso-butyric and n-valeric acids, L-lactic acid and D-lactic acid, etc) among infants receiving an investigational formula, infants receiving a control formula, and breastfeeding infants.

ELIGIBILITY:
Inclusion Criteria:

* 10-14 days of age at enrolment and randomization, inclusive (day of birth is considered day 0)
* Plan to exclusively formula feed (formula groups) OR exclusively feed human milk (breastfeeding group)
* Healthy singleton birth
* Gestational age of 37-42 completed weeks (37 weeks 0 days through 42 weeks 6 days)
* Birth weight of 2490g to 4200g
* Signed informed consent obtained for infant's and mother's participation in the study

Exclusion Criteria:

* History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the Investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant
* Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake, at time of randomization (at investigator discretion)
* Known allergy to cow's milk protein or a well-documented family history of allergy to cow's milk protein
* Weight at randomization is <90% of birth weight [(weight at Visit 1÷birth weight) x 100 <90%]
* Immunocompromised (according to a doctor's diagnosis of immunodeficiency such as Combined Immunodeficiencies, DiGeorge Syndrome, Wiskott-Aldrich Syndrome, Severe Congenital Neutropenia and Secondary Immunodeficiencies linked to HIV infection, Down Syndrome or others)
* Known head/brain disease/injury such as microcephaly, macrocephaly or others.
* Enrollment in another interventional clinical research study while participating in this study

Ages: 10 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of change in body weight (grams/day) from baseline | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks
  Rate of change in body weight (grams/day) between baseline and B+2 weeks, B+4 weeks, B+8 weeks, B+12 weeks, and B+16 weeks.

SECONDARY OUTCOMES:
Rate of change in body length (mm/day) from baseline | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks
  Rate of change in length (mm/day) measured between baseline (B) and B+2 weeks, B+4 weeks, B+8 weeks, B+12 weeks, and B+16 weeks.
Rate of change in head circumference (mm/day) from baseline | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks
  Rate of change in head circumference (mm/day) measured between baseline (B) and B+2 weeks, B+4 weeks, B+8 weeks, B+12 weeks, and B+16 weeks.
Achieved body weight | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks
  Achieved body weight (grams) at each study visit
Achieved body length | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks
  Achieved body length (cm) at each study visit
Achieved head circumference | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks
  Achieved head circumference (cm) at each study visit
Percentages of infants in each group who are <10th percentile in weight for age. | 16 weeks
  Percentages of infants in each group who are <10th percentile in weight for age.
Percentages of infants in each group who are <10th percentile in length for age. | 16 weeks
  Percentages of infants in each group who are <10th percentile in length for age.
Percentages of infants in each group who are <10th percentile in head circumference for age. | 16 weeks
  Percentages of infants in each group who are <10th percentile in head circumference for age.
Adverse events rate | 16 weeks
  Number and percentages of infants in each group experiencing any adverse events and any serious adverse events
Average daily formula intake | 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks
  Average daily formula intake volume based on 3-day records kept by parents or care-givers prior to each study visit.
Percentage of fussiness | 16 weeks
  Percentages of parents in each group reporting fussiness
Percentage of colic | 16 weeks
  Percentages of parents in each group reporting colic
Percentage of patterns | 16 weeks
  Percentages of parents in each group reporting sleeping patterns
Percentage of cramps | 16 weeks
  Percentages of parents in each group reporting cramps
Percentage of regurgitation | 16 weeks
  Percentages of parents in each group reporting regurgitation
Stool characteristics | 16 weeks
  Score of stool characteristics
Percentage of respiratory manifestations | 16 weeks
  Percentages of parents in each group reporting respiratory manifestations
Percentage of dermatologic manifestations | 16 weeks
  Percentages of parents in each group reporting dermatologic manifestations
Fecal Bifidobacteria counts | 8 weeks,16 weeks
  Total fecal Bifidobacteria counts (mean log10 counts / g wet-weight stool) at 8 weeks and 16 weeks.
Fecal Lactobacillus counts | 8 weeks,16 weeks
  Total fecal Lactobacillus counts (mean log10 counts / g wet-weight stool) at 8 weeks and 16 weeks.
Stool short-chain fatty acid | 8 weeks,16 weeks
  Total stool short-chain fatty acid metabolites in mg/g dry stool at 8 weeks and 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - Jinhua Nanyuan Community Health Center (site 1919), Jinhua, Zhejiang
  - Jinhua Qiubin Community Health Center (site 1969), Jinhua, Zhejiang
  - Jinhua Xiguan Community Health Center (site 1966), Jinhua, Zhejiang